CLINICAL TRIAL: NCT04423328
Title: Assistant Head Nurse (Department of Nursing, Taipei Veterans General Hospital, Taipei, Taiwan)
Brief Title: Establishment of Sleep Quality, Physical and Mental Health and Occupational Burnout Management Model for Shift Nursing Staff and Evaluation of Its Effectiveness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-03-014BC
Record Dates: First submitted 2020-05-27; First posted 2020-06-09 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Sleep Quality; Occupational Burnout
Keywords: Sleep disturbances; HRV monitoring watch; health status; shift rotation nurses; Occupational Burnout; acupressure
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Burnout, Professional; Parasomnias | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure (Experimental): Every day before going to sleep, massage acupoints for eight consecutive weeks, followed by Shenmen→Neiguan→Hegu acupoints.
  Interventions: Behavioral: acupressure
- sham acupressure (Sham Comparator): Every day before going to sleep, massage acupoints for eight consecutive weeks, followed by Waiguan→Liangqiu→Tiaokou→ Chengshan acupoints
  Interventions: Behavioral: acupressure

INTERVENTIONS:
Behavioral: acupressure — self-acupressure

SUMMARY:
The purpose of this study was to investigate the relationship between the personal characteristics and work characteristics of shift nurses and occupational burnout, sleep quality and physical and mental health. Use " acupressure " as an intervention to compare the status of shift nurses before and after intervention and to track after interventional therapy, 1, 2, and 3 months of longitudinal results.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the relationship between the personal characteristics and work characteristics of shift nurses and occupational burnout, sleep quality and physical and mental health. Use " acupressure " as an intervention to compare the status of shift nurses before and after intervention and to track after interventional therapy, 1, 2, and 3 months of longitudinal results. Use the "Smart Care VIP bracelet" to detect physical and mental conditions (psychological stress, physical fatigue) to assess the applicability of the Smart Care VIP bracelet as a "Shift Care Staff Sleep Quality, Physical and Mental Health and Occupational Burnout Management System" and evaluate effectiveness, and establishment of an effective management system.

Most studies in China have shown that the use of acupressure to improve the sleep quality of nursing staff generally has its efficacy, but the lack of research at proves that acupressure is used by nursing staff to improve sleep quality and improve occupational burnout. It is expected to be from May to December 2020. The nursing staff of a medical center in Taipei will be selected for stratified sampling. The conditions for receiving the case are shift nurses who have served in the institution for more than one year. Subjective sleep is assessed using Epworth sleepiness scale. The objective part is to use the "Smart Care VIP Bracelet" to measure sleep time; Chinese version of the Chinese Health Questionnaire-12 (CHQ-12) and occupational burnout scale questionnaire as a tool for discussion. It is planned to randomly assign shift nurses to 42 acupressure groups and control group (sham), and use activity record (Smart Care VIP bracelet) to monitor and record fatigue Index and stress changes.

ELIGIBILITY:
Inclusion Criteria:

1. Shift nursing staff who have been employed in this institution for more than one year, and there have been more than two shift types in the past year. Can fill out the questionnaire and agree to participate in this research and sign the consent form.
2. Chinese Health Questionnaire-12 > 1.5
3. Epworth sleepiness scale > 6.5 points

Exclusion Criteria:

1. Long-term (more than one month) taking sleeping pills such as Benzodiazepines, Stilnox, Imovane, etc.
2. Nursing staff in the same ward as the PI.
3. Encountered major life problems one month before the intervention, such as: falling out of love, family member's accident, personal diagnosis of illness, etc.

Ages: 22 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-08-28 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
sleep quality | 3 months
  Epworth sleepiness scale(ESS)Epworth sleepiness Scale - Taiwan form (ESS-T):
  .The internal consistency of the scale Cronbach's α = .81, and then measured the reliability r = .74, p = .001.
  .The evaluation of the degree of drowsiness is expressed as a score of zero (never occurred) to three (almost all), with a total of 24 points.
  The higher the total score, the more severe the level of drowsiness. A zero score indicates the best situation.
Physical and Mental Health | 3 months
  Chinese Health Questionnaire-12 (CHQ-12):
  The reliability and validity of Cronbach'α was 0.83-0.92 (Cheng et al., 1990) CHQ-12 has 12 questions in total, two of which are positive. Ten questions of which are negative. It is a self-reported four-point scale. It is score from 0-0-1-1, with a total score of 12 points.
Chinese version of the Occupational Burnout Inventory: | 3 months
  The occupational burnout inventory consists of four subscales with 21 questions.
  All subscales have a score range of 0-100 points. The scale is measured by the respondent self-assessed the frequency of various problems in the past week.
  The total scale score is the sum of all subscale scores, and the higher the score, the higher the worker's feeling of burnout.
  The four subscales in the scale include personal burnout (5 questions), work burnout (5 questions), overwork (5 questions) and client burnout (6 questions).
  The Cronbach'α of the scale is above 0.84, and the scale has good construction validity and standard validity (Chang et al., 2007; Tseng, & Cheng, 2002; Yeh, Cheng, Chen, & Chiu, 2008).

SECONDARY OUTCOMES:
Heart Rate Variability, HRV -「Smart Care VIP Bracelet Watch」 | 3 months
  The "Smart Care VIP Bracelet Watch" worn on the subject's wrist for HRV monitoring to record changes in the individual's physical activity.
  The contents of the record include the total daily sleep time (hours), waking time (minutes), number of waking, physical and mental index (mental stress, physical burnout) and other data for each case.
  To obtain the heart rate variability index directly, which represents the low frequency (LF) (%) of the sympathetic nerve activity index.
  High frequency power (HF) (%) representing the parasympathetic nerve activity index, and low frequency / high frequency power ratio (LF / HF) representing the sympathetic / parasympathetic balance index.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shan Jan, master, Principal Investigator — Department of Nursing, Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Department of Nursing, Taipei Veterans General Hospital,, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng TA, Wu JT, Chong MY, Williams P. Internal consistency and factor structure of the Chinese Health Questionnaire. Acta Psychiatr Scand. 1990 Oct;82(4):304-8. doi: 10.1111/j.1600-0447.1990.tb01389.x. PMID 2260484
- [Background] Chang, Y.J., Yeh, W.Y., Chen, C.W., Chen, C.J., Shih, T.S., & Cheng, Y.W. (2007). Distribution and Correlates of Burnout among Paid Employees in Taiwan. Taiwan Journal of Public Health, 26(1), 75-87. doi:10.6288/TJPH2007-26-01-09
- [Background] Tseng, H.P., & Cheng, Y.W. (2002). Reliability and Validity of the Chinese Demand-Control-Support Model and Effort-Reward Imbalance Model Questionnaires: a Study Among Employees of the Microelectronic Industry. Taiwan Journal of Public Health, 21(6), 420-432. doi:10.6288/TJPH2002-21-06-05
- [Background] Yeh, W.Y., Cheng, Y.W., Chen, M.J., & Chiu, W.H. (2008). Development and validation of an occupational burnout inventory. Taiwan Journal of Public Health, 27(5), 349-364. doi: 10.6288/TJPH2008-27-05-01